CLINICAL TRIAL: NCT06584630
Title: Molecular Classification of Endometrial Cancer: Impact on Adjuvant Treatment Planning.
Status: Active, not recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Dimitrios Zouzoulas, Dr, Aristotle University Of Thessaloniki
Other Study IDs: 37577
Record Dates: First submitted 2024-07-04; First posted 2024-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- endometrial cancer patients that underwent molecular classification

SUMMARY:
Molecular classification that has been recently incorporated in FIGO classification of endometrial cancer is a new triage tool for the better management of endometrial cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of endometrial cancer.
* Surgical treatment at our Gynecological - Oncology Unit.

Exclusion Criteria:

* Refusal to be tested for the molecular classification
* Presence of a synchronous neoplasm.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Endometrial cancer patients that underwent surgery and were tested for molecular analysis (POLE, MSI, p53)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Multidisciplinary Team Board decision change | 2 years (study completion)
  MDT decision for adjuvant treatment (Rate of adjuvant treatment change)

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Department of Obstetrics & Gynecology, AUTh, "Papageorgiou" Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No